CLINICAL TRIAL: NCT03843996
Title: Comparison of a Novel Wound Dressing Stratamed Versus Current Clinical Practice After Follicular Unit Extraction Hair Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stratpharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: SPASM06
Record Dates: First submitted 2019-02-11; First posted 2019-02-18 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Wounds and Injuries
Keywords: Stratamed; wound healing; follicular unit extraction hair transplantation
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: This Phase IV, post-marketing, single center study will be a single-blind, within subject split scalp efficacy comparison of Stratamed® and standard clinical practice, Bacitracin, post FUE. Twenty subjects desiring to undergo FUE for hair restoration will apply Stratamed® on one half of the donor area on the back of the scalp and Bacitracin on the other side at least twice a day for a week post procedure. The side of the scalp receiving each product will be randomized, and the evaluating physician will be blinded. Subjects will be evaluated, photographed, and will fill out subject reported questionnaires live at days 1 (+1) and 7 (±1) post procedure. Subjects will also fill out the subject reported questionnaires at home in between live study visits (days 2, 3, 4, 5, and 6).
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: This is an randomized, single-blind, split-scalp study, such that subjects will know what side of the scalp the investigational and standard treatment products are applied. The PI will evaluate efficacy and safety blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment left (Experimental): A randomized side of the scalp will be treated with Stratamed®, the other side with standard clinical practice.
  Interventions: Device: Treatment - Stratamed
- Treatment right (Experimental): A randomized side of the scalp will be treated with Stratamed®, the other side with standard clinical practice.
  Interventions: Device: Treatment - Stratamed

INTERVENTIONS:
Device: Treatment - Stratamed — To determine if Stratamed is more effective than standard of care therapy in limiting severity and duration of signs and symptoms of acute inflammation post follicular harvesting procedure.
  Other Names: wound healing

SUMMARY:
Follicular donor sites on the scalp for hair transplantation will be treated with studied products post harvest.

A randomized side of the scalp will be treated with Stratamed, the other side with standard clinical practice.

Subjects will be assessed live immediately post treatment and in 2 sessions during the healing phase post harvest. Subjects will also complete subject reported outcome questionnaires at home between study visits.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Able to provide informed consent
* Planning to undergo follicular unit extraction hair restoration

Exclusion Criteria:

* Significant medical or surgical conditions
* Unable to give informed consent
* Patient unable to apply topical device
* Allergy or intolerance to ingredients or excipients of the formulation of studied products
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2019-01-08 (Actual)

PRIMARY OUTCOMES:
Wound healing change over time from day 0 to day +1 (+1), to day +7 (±1) | duration of the studybe evaluated and rated on days 1 (+1) and 7 (±1) post procedure for both the investigational and standard treatment products
  Stratamed will improve the healing response vs. current standard of care therapy. Healing Response (4 point ordinal scale)
  LEFT SIDE
  * Not healed at all (0%)
  * Mildly healed (33%)
  * Moderately healed (66%)
  * Completely healed (100%)
  RIGHT SIDE
  * Not healed at all (0%)
  * Mild healing (33%)
  * Moderately healed (66%)
  * Completely healed (100%)

CONTACTS AND LOCATIONS:
Locations (1):
- New Jersey Plastic Surgery, Montclair, NJ USA, Montclair, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
all IPD that underlie results for a publication